CLINICAL TRIAL: NCT04957862
Title: Robotic Assisted Evacuation of Subacute and Chronic Supratentorial Deep Hypertensive Intracerebral Hemorrhage for Accelerating Functional Rehabilitation (RESCUE-CHAIN): a Multi-center Randomized Controlled Trial
Brief Title: Robotic Assisted Evacuation of Subacute and Chronic Supratentorial Deep Hypertensive Intracerebral Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Beijing Tian Tan Hospital Affiliated to Capital Medical University (Unknown); Tianjin Medical University General Hospital (Other); Peking Union Medical College Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Renmin Hospital of Wuhan University (Other); South Taihu Hospital of Huzhou (Unknown); Qian Xi Nan People's Hospital (Unknown); Huazhong University of Science and Technology Union Hospital (Nanshan Hospital) (Unknown); Fujian Provincial Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); LanZhou University (Other); Anhui No.2 Provincial People's Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Jinjiang Hospital of Traditional Chinese Medicine (Unknown); Tang-Du Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shenzhen People's Hospital (Other); Shaanxi Provincial People's Hospital (Other); Shanghai 6th People's Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Sanhe Yanjiao People's Hospital (Unknown); General Hospital of Ningxia Medical University (Other); Affiliated Hospital of Chifeng University (Unknown); Haikou People's Hospital (Other); Qilu Hospital of Shandong University (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Hou Lijun, Professor, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE-CHAIN
Record Dates: First submitted 2021-07-03; First posted 2021-07-12 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hypertensive Intracerebral Hemorrhage
Keywords: Randomized controlled trial; Hypertensive Intracerebral Hemorrhage; subacute; chronic; robotic assisted evacuation; function rehabilitation
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robotic assisted evacuation (Active Comparator): In the intervention arm, patients will receive stereotactic robotic assisted HICH evacuation according to the protocol under general anesthesia.
  Interventions: Procedure: Robotic Assisted Evacuation
- Concomitant care (No Intervention): All enrolled HICH patients in this study will receive standard medical treatment in the first 3-4 weeks according to the ASA/AHA guideline . Continued medical treatment is applied to patients in the control arm. Both arms will receive identical rehabilitation therapy three times per week for 180 days at one facility. Rehabilitation therapy includes identical physical therapy, occupational therapy, speech therapy, functional training, acupuncture and massage.

INTERVENTIONS:
Procedure: Robotic Assisted Evacuation — On the day of surgery, the patient is placed in the prone position. After the Mayfield skull clamp is positioned to reduce interference, the videometric tracker of robot will automatically scan the preliminary markers to complete patient-to-image registration. Following the registration, the robotic arm will move on command according to the planned puncture trajectory and stop at a defined distance to the marked target point. The entry point is marked on the scalp along the puncture trajectory, then a scalp incision and burr-hole drilling will be performed. After penetrating the dura with unipolar electrocautery, a drainage tube will be gently inserted to the defined depth under the indication of the disinfected robotic arm. The liquefied hematoma will be withdrawn slowly by a 10 mL syringe.
  Arms: robotic assisted evacuation

SUMMARY:
Robotic Assisted Evacuation of Subacute and Chronic Supratentorial Deep Hypertensive Intracerebral Hemorrhage for Accelerating Functional Rehabilitation (RESCUE-CHAIN): a Multi-center Randomized Controlled Trial

DETAILED DESCRIPTION:
Background: Hypertensive intracerebral hemorrhage (HICH) is a devastating neurological disorder with high mortality and disability rates. Secondary injury following HICH may worsen motor function rehabilitation in subacute and chronic hematoma. Hematoma evacuation has the potential to reduce mass effect and mitigate the neurotoxic effects. A per-protocol analysis identified a significant functional improvement in patients with minimally invasive surgery with thrombolysis achieving end of treatment (EOT) goal ≤ 15mL. However, no surgical management of stabilized subacute or chronic HICH have been reported before. Therefore, we design this study in which we hypothesize this robotic assisted approach to hematoma EOT goal ≤ 15mL would accelerate functional rehabilitation in subacute and chronic HICH patients.

ELIGIBILITY:
The inclusion criteria are HICH patients who: (1) are ≥ 18 and ≤ 75 years old of either gender; (2) have evidence of supratentorial, deep-seated on CT scan with a volume of between 15 mL and 30 mL; (3) are within 24 h of ictus (<24 h between symptom onset and initial imaging); (4) have stable hematoma (hematoma growth<5 mL) for at least 12 h after diagnostic CT; (5) have no brain herniation and no needs for emergency surgery (clinical decisions made by 2 attending neurosurgeons); (6) have had no previous surgery on HICH or traumatic brain injury; (7) have GCS>8, NIH Stroke Scale (NIHSS)>5, Modified Rankin Scale (mRS) 3-5, and FMA scale<85; (8) fully understand the nature of the study and have signed informed consent.

The exclusion criteria are: (1) HICH caused by aneurysms, cerebrovascular malformations, tumors or trauma; (2) any pre-existing physical or mental disorder that could interfere with the functional assessment; (3) severe abnormal coagulation function, hematologic diseases or multiple hemorrhagic lesions; (4) excessive hematoma extending into the ventricular system with ventricular dilation; (5) concomitant diseases such as liver, kidney and heart failure; (6) rebleeding>5 mL or with surgical indications before allocation; (7) poor adherence or other unsuitable situations for the trial as determined by the investigators; (8) pregnant female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) 0-2 | 180 days after surgery
  The modified Rankin Scale (mRS) is a single item, global outcomes rating scale for patients post-stroke. It is used to categorize level of functional independence with reference to pre-stroke activities rather than on observed performance of a specific task.

SECONDARY OUTCOMES:
Evacuation rate of HICH | at the first day after procedure, 30 days and 180 days during the follow-up period.
  the ratio of effective volume reduction to the initial volume
modified Rankin Scale (mRS) 0-1 | 180 days after surgery
  The modified Rankin Scale (mRS) is a single item, global outcomes rating scale for patients post-stroke. It is used to categorize level of functional independence with reference to pre-stroke activities rather than on observed performance of a specific task.
between-group shift analysis in the mRS distribution | 180 days after surgery
  The modified Rankin Scale (mRS) is a single item, global outcomes rating scale for patients post-stroke. It is used to categorize level of functional independence with reference to pre-stroke activities rather than on observed performance of a specific task.
Extended Glasgow Outcome Scale (eGOS) | at 90- and 180-days after surgery.
  The GOS-E adds to the original 5 GOS categories, with 3 additional categories. The 8 categories are: Dead, Vegetative State, Lower Severe Disability, Upper Severe Disability, Lower Moderate Disability, Upper Moderate Disability, Lower Good Recovery, and Upper Good Recovery.
NIH Stroke Scale（NIHSS） | at 90- and 180-days after surgery.
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The single patient assessment requires less than 10 minutes to complete. The evaluation of stroke severity depends upon the ability of the observer to accurately and consistently assess the patient
Barthel Index for Activities of Daily Living (ADL-BI) | at 90- and 180-days after surgery.
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. The index also indicates the need for assistance in care.
Fugl-Meyer Assessment (FMA) | at 90- and 180-days after surgery.
  The FMA motor assessments for the upper (maximum score 66 points) and lower extremity (maximum score 34 points) are recommended as core measures to be used in every stroke recovery and rehabilitation trial.
Motor Assessment Scale (MAS) | at 90- and 180-days after surgery.
  The MAS is comprised of 8 items corresponding to 8 areas of motor function. Patients perform each task 3 times and the best performance is recorded.
  Supine to side lying Supine to sitting over the edge of a bed Balanced sitting Sitting to standing Walking Upper-arm function Hand movements Advanced hand activities

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Hou, MD,PhD, Principal Investigator — Shanghai Changzheng Hospital; Tao Xu, MD,PhD, Study Director — Shanghai Changzheng Hospital

IPD SHARING:
Plan to Share IPD: No